CLINICAL TRIAL: NCT01289756
Title: Influence of Pharmacogenetic Factors, Paroxetine and Clarithromycin on Pharmacokinetics of Clomiphene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Responsible Party: Principal Investigator, Matthias Schwab, Prof. M.D., Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IKP237; 2009-014531-20 (EudraCT Number)
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Anovulation; Disorder Due Cytochrome P450 CYP2D6 Variant; Cytochrome P450 CYP3A Enzyme Deficiency
Keywords: pharmacokinetic; clomiphene; CYP2D6 polymorphisms; inhibition of CYP2D6 and CYP3A4
MeSH Terms: conditions — Anovulation | interventions — Clomiphene; Paroxetine; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CYP2D6 EM (Experimental): clomiphene, clomiphene and paroxetine, clomiphene and clarithromycin
  Interventions: Drug: Clomiphene; Drug: clomiphene and paroxetine; Drug: clomiphene and clarithromycin
- CYP2D6 IM (Experimental): clomiphene, clomiphene and paroxetine, clomiphene and clarithromycin
  Interventions: Drug: Clomiphene; Drug: clomiphene and paroxetine; Drug: clomiphene and clarithromycin
- CYP2D6 PM (Experimental): clomiphene, clomiphene and paroxetine, clomiphene and clarithromycin
  Interventions: Drug: Clomiphene; Drug: clomiphene and paroxetine; Drug: clomiphene and clarithromycin
- CYP2D6 UM (Experimental): clomiphene, clomiphene and paroxetine, clomiphene and clarithromycin
  Interventions: Drug: Clomiphene; Drug: clomiphene and paroxetine; Drug: clomiphene and clarithromycin

INTERVENTIONS:
Drug: Clomiphene — clomiphene once 100 mg oral
Drug: clomiphene and paroxetine — clomiphene 100mg and paroxetine 3x40mg
Drug: clomiphene and clarithromycin — clomiphene 100mg and clarithromycin 9x500mg

SUMMARY:
Aim of the study is the clinical validation of the metabolism and the pharmakokinetic of Clomifen in correlation to CYP2D6 and inhibition of CYP3A4.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Female caucasians
* Age 18 - 45 years old
* BMI 18.5 - 26 kg/m2

Exclusion Criteria:

* Persons with known sensitivity of Clomifen and/or Paroxetine and/or Clarithromycin
* Pregnancy/lactation period
* Meno-/postmenopausal
* Smokers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC)of clomiphene | 1, 2, 4, 6, 8, 10, 12, 24, 72 and 168 hours after durg application
  AUC of clomiphene and metabolites
Peak Plasma Concentration (Cmax)of Clomiphene | 1, 2, 4, 6, 8, 10, 12, 24, 72 and 168 hours after drug application
  Cmax of Clomiphene and metabolites

SECONDARY OUTCOMES:
Clearance of Clomiphene | 4, 8, 12 and 24 hours after drug application
  Clearance of Clomiphene and metabolites
Metabolomic | 4, 8, 12 and 24 hours after drug application
  Metabolomic
Tmax of clomiphene | 4, 8, 12, 24 hours after drug application
  Tmax of clomiphene and metabolites
Pharmacogenomics | once
  Pharmacogenomics

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Schwab, Prof., Principal Investigator — Dr. Margarete Fischer-Bosch-Institute of Clinical Pharmacology
Locations (1):
- Dr. Margarete Fischer-Bosch-Institute of Clinical Pharmacology and University of Tuebingen, Stuttgart, Baden-Wurttemberg, Germany